CLINICAL TRIAL: NCT04242719
Title: Management of Deep Retinal Capillary Ischemia by Electromagnetic Stimulation and Platelet- Rich Plasma
Acronym: rEMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Universitesi Teknokent (Other)
Responsible Party: Principal Investigator, Umut Arslan, Principle investigator, MD, Ankara Universitesi Teknokent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-1177-18
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Deep Retinal Capillary Ischemia; Paracentral Acute Middle Maculopathy; Acute Macular Neuroretinopathy
Keywords: Deep retinal capillary ischemia; Paracentral acute middle maculopathy; Acute macular neuroretinopathy; Electromagnetic stimulation; Magnovision; Platelet-rich plasma
MeSH Terms: conditions — White Dot Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, comparative
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Only electromagnetic stimulation (Active Comparator): Only rEMS was preferred as the initial step
  Interventions: Device: Electromagnetic stimulation
- Combined with electromagnetic stimulation and PRP (Active Comparator): Order to augment the effect of the rEMS, sub-tenon aPRP injection was added.
  Interventions: Device: Electromagnetic stimulation; Biological: Platelet rich plasma
- Natural course (No Intervention): Served as control group, and existing systemic disorder(s) were consulted and treated accordingly.

INTERVENTIONS:
Device: Electromagnetic stimulation — Retinal electromagnetic stimulation A high-frequency repetitive electromagnetic stimulation protocol has been defined in the literature and was applied in groups 1 and group 2 via a novel device developed specifically for ophthalmic usage (Magnovision-TM, Bioretina Biyoteknoloji AŞ, Ankara,Turkey). The patients underwent 10 consecutive sessions of rEMS application. Parameters for the treatment were 42 hertz frequency/min, 30 minutes of duration and mild operating cycle. The power of the electromagnetic field was 2000 milligauss, which is a very low dose and within the safety limits of World Health Organisation. In group 2, sub-tenon aPRP injections were also performed immediately after the first, fifth, and tenth sessions of rEMS application.
  Other Names: Magnovision
  Arms: Combined with electromagnetic stimulation and PRP; Only electromagnetic stimulation
Biological: Platelet rich plasma — About 20 ml of blood was drawn from the patient's antecubital vein and inserted into two 10-ml vacutainer tubes that contain trisodium citrate (T-LAB PRP Kit, T-Biyoteknoloji, Bursa, TURKEY). These tubes were placed in a refrigerated (+4 °C) centrifuge (Nüve NF 1200R, Nüve Laboratuar Teknolojileri, Ankara, TURKEY) and spun at 2500 rpm (580×g) for 8 min within 30 min of collection. Three different layers formed in the tubes: red blood cells at the bottom, platelet-rich plasma in the middle, and platelet-poor plasma in the top layer. A total of 1.5 ml of the middle layer (which mainly contained platelets) was withdrawn by syringe and immediately injected into the sub-tenon space of each eye after topical anesthesia with proparacaine hydrochloride (Alcaine, Alcon, USA) drops.
  Other Names: Autologous PRP
  Arms: Combined with electromagnetic stimulation and PRP

SUMMARY:
To investigate the efficacy of retinal electromagnetic stimulation and sub-tenon autologous platelet rich plasma in the treatment of deep retinal capillary ischemia.

DETAILED DESCRIPTION:
Deep retinal capillary ischemia (DRCI) is a recently described entity in patients presenting with an acute-onset paracentral scotoma. Subclinical macular lesions of DRCI were formerly best visualized on near-infrared reflectance imaging. The development of optical coherence tomography angiography (OCTA) has facilitated studies of the retinal capillary structures. The multiplanar superficial capillary plexus is located in the inner plexiform layer (IPL) and contains synapses between bipolar and ganglion cells as well as amacrine cells. The deep capillary plexus (DCP) is located in the outer plexiform layer (OPL), which is thinner than the IPL. The DCP is composed of synapses of photoreceptors, bipolar cells, and horizontal cells. This area is also at the border of the oxygen diffusion from the choroid. It is likely that the oxygen coming from the choroid has been completely consumed by the photoreceptors because of the low partial pressure of oxygen level in the outer nuclear layer (ONL). The DCP supplies both the bipolar cells and the synaptic structure of the OPL and Henle ﬁbers.

Deep retinal capillary ischemia is an ischemic event in the middle and deep layers of the retina due to various systemic or local vascular pathologies. It is obvious in the intraretinal hyper-reflective bandlike zone located superior or inferior to the OPL conjointly on in a structural cross-sectional B-scan of the spectral domain optical coherence tomography (SD-OCT) examination along with an acute-onset paracentral scotoma and subjective complaints of the patient. Ophthalmologists often face a significant diagnostic challenge because of a lack of noticeable changes in the appearance of the retina.

DRCI has two different appearances on B-scan SD-OCT exams according to the level of the involved DCP. If the hyper-reflective bandlike zone is located on the outer plexiform layer-inner nuclear layer (OPL-INL) junction, then it is termed "Paracentral Acute Middle Maculopathy (PAMM)" or type-1 deep retinal capillary ischemia. If the hyper-reflective band is seen on the OPL-ONL junction, then it is termed as type-2 deep retinal capillary ischemia. This might be a new variant of "Acute Macular Neuroretinopathy (AMN)". These intraretinal hyperreflective zones are seen as patchy areas of various patterns on en-face OCT image, and atrophic areas in the inner and the outer nuclear layer respectively are developed in the late stage of the diseases. The pathophysiologic features of DCP ischemia is considered to be ischemic hypoxia leading to cell death with swelling of the middle retinal tissues. This may lead to severe vision loss and permanent paracentral scotoma depending on the underlying cause and depth of ischemia. It can also be observed by slowing metabolic activity in photoreceptors and neural retina. The metabolic slowdown is defined as a dormant phase in photoreceptors and OFF mode in the neural retina.

The retinal deep capillary plexus is a single monoplanar capillary plexus located in the OPL. It has the lowest vessel density-this is a signiﬁcant ﬁnding that might be used to evaluate retinal vascular diseases accurately. For this reason, the changes in the percentage of the vessel density in DCP during the follow-up were preferred as an assessment parameter of the treatment modalities used in this prospective clinical study.

Platelets are anucleated cells that contain many types of growth factors including platelet-derived growth factor(PDGF), transforming growth factor-β(TGF-β), vascular endothelial growth factor(VEGF), and epidermal growth factor(EGF) in alpha granules. Thus, the supplementation of growth medium with autologous platelet-rich plasma (aPRP) could be desirable for clinical applications and could lead to some functional improvement.

High-frequency repetitive electromagnetic stimulation (rEMS) has promising therapeutic potential in ischemic neurological patients. The rationale of rEMS is that it modulates neural excitability and increases neural plasticity; thus, it improves the functional outcome. These neuroprotective effects of rEMS are dependent on the increase in the level of brain-derived neurotrophic factor (BDNF), VEGF, and increased tyrosine kinase A, B, and C (TrkA, TrkB, and TrkC) receptor activation. Therefore, high-frequency rEMS might be a promising therapeutic strategy for ischemic retinal disorders such as DRCI.

There is no known and proven specific treatment for DRCI to date except for systemic check-ups and treatment of the underlying diseases or predisposing factors. The aim of this preliminary clinical study is to investigate the efficacy of high-frequency rEMS alone or in combination with sub-tenon fresh aPRP as a treatment modality in the treatment of DRCI. To the best of our knowledge, this is the first prospective clinical trial on this subject in the ophthalmic literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining of blurred vision and/or acute-onset paracentral scotoma during the last month without any visible fundus change along with typical SD-OCT and OCTA findings.

Exclusion Criteria:

* The presence of noticeable changes in the fundus examination,
* Any optic media opacity that may cause artefacts on OCTA images and interfere with quantitative measurements of the DCP vessel density,
* Complaining of paracentral scotoma lasting more than 1 month (in order to exclude chronic changes in the retinal tissue),
* Presence of atrophic changes in INL or ONL on cross-sectional B-scan SD-OCT

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Deep retinal capillary vessel density | Change from baseline deep reinal capillary vessel density at 1 month.
  The vessel densities (in %) of deep capillary plexus were measured with "AngioAnalytic" feature of the OCTA device. To compare the percentage of the vessel densities precisely during follow-up, the "Link-B Scans" button on the screen was activated so that the exact same segmentation planes of the DCP could be compared. The OCTA device automatically calculated and displayed the vessel density maps as follow-up sequences (Angio Retina multiscan view) and trend analysis.
Best corrected visual acuity | Change from baseline best corrected visual acuity at 1 month.
  Number of readable letters after glasses correction

CONTACTS AND LOCATIONS:
Overall Officials: Umut Arslan, MD, Principal Investigator — Ankara Universitesi Teknokent
Locations (1):
- Ankara University Biotechnology Institute, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nemiroff J, Kuehlewein L, Rahimy E, Tsui I, Doshi R, Gaudric A, Gorin MB, Sadda S, Sarraf D. Assessing Deep Retinal Capillary Ischemia in Paracentral Acute Middle Maculopathy by Optical Coherence Tomography Angiography. Am J Ophthalmol. 2016 Feb;162:121-132.e1. doi: 10.1016/j.ajo.2015.10.026. Epub 2015 Nov 10. PMID 26562176
- [Background] Arslan U, Ozmert E, Demirel S, Ornek F, Sermet F. Effects of subtenon-injected autologous platelet-rich plasma on visual functions in eyes with retinitis pigmentosa: preliminary clinical results. Graefes Arch Clin Exp Ophthalmol. 2018 May;256(5):893-908. doi: 10.1007/s00417-018-3953-5. Epub 2018 Mar 15. PMID 29546474
- [Background] Luo J, Zheng H, Zhang L, Zhang Q, Li L, Pei Z, Hu X. High-Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) Improves Functional Recovery by Enhancing Neurogenesis and Activating BDNF/TrkB Signaling in Ischemic Rats. Int J Mol Sci. 2017 Feb 20;18(2):455. doi: 10.3390/ijms18020455. PMID 28230741
- [Result] Ozmert E, Arslan U. Management of Deep Retinal Capillary Ischemia by Electromagnetic Stimulation and Platelet-Rich Plasma: Preliminary Clinical Results. Adv Ther. 2019 Sep;36(9):2273-2286. doi: 10.1007/s12325-019-01040-2. Epub 2019 Aug 5. PMID 31385285